CLINICAL TRIAL: NCT05908669
Title: Deuterium Metabolic Imaging to Assess Radiotherapy Changes in Glioblastoma Multiforme
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DMI-GBM
Record Dates: First submitted 2023-05-15; First posted 2023-06-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GBM patients, IDH-wt
  Interventions: Diagnostic Test: Deuterium metabolic imaging

INTERVENTIONS:
Diagnostic Test: Deuterium metabolic imaging — MRI after oral administration of 75g of [6,6'-2H2]glucose.

SUMMARY:
This is a feasibility single arm study designed for obtaining early data for optimization and evaluation of the clinical potential for a new MR technique using deuterated glucose. The purpose of the study is to investigate whether this technique is useful in metabolic imaging of glioblastoma multiforme (GBM) and whether radiochemotherapy (RCT) induced changes in the brain metabolism can be detected and might be predictive for treatment response. The study will include 10 patients with histologically verified GBM scheduled for standard RCT. Patients will have MRI scan performed before and within 8 weeks after starting RCT. The scans will include imaging after oral intake of deuterated glucose, so called deuterium metabolic imaging (DMI). Based on this study, the most optimal scanning technique, output variables of highest discriminative power with respect to RCT, and potential predictive markers for response will be selected for further clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed GBM IDHwt
* Scheduled for long-course radiotherapy
* At least 18 years of age
* WHO performance status 0-1
* Women who are not postmenopausal or surgically sterile must have a negative serum or urine pregnancy test performed at time of inclusion in the study. Safe and highly effective contraception must be used throughout the study meaning either hormonal anti-conception or an anti-fertility intrauterine device.
* Danish speaking
* Able and willing to comply after informed consent

Exclusion Criteria:

* Subjects who are receiving any other investigational agents.
* Previous or current treatment by radiation or chemotherapy.
* History of alcohol abuse or illicit drug use.
* Contraindications to MRI Pacemaker, neurostimulator or cochlea implant Metal foreign bodies such as fragments and irremovable piercings Unsafe medical implants Intracranial clips or coils Claustrophobia Largest circumference including arms > 160 cm
* Contraindications to gadolinium contrast eGFR ≤ 30 mL/min/1.73m2 Previous adverse reactions to gadolinium
* Not able or willing to receive radiotherapy
* Predicted remaining survival <3 months
* Insulin-treated diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed GBM, idh-wt (performance 0-1) are enrolled before initiating radiochemotherapy. They are not allowed to have contraindications to MRI with contrast or diabetes.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Deuterium Metabolic Imaging | Imaging repeated twice with ~10 weeks between them.
  2H-glucose uptake and conversion to lactate and glx over 120 minutes in normal brain and tumor tissue. Before and after radiochemotherapy to measure the changes with therapy.

SECONDARY OUTCOMES:
Perfusion MRI | Imaging repeated twice with ~10 weeks between them.
  Dynamic contrast enhancement MRI using a gadolinium-based contrast agent.
Microvascular diffusion MRI | Imaging repeated twice with ~10 weeks between them.
  Diffusion-weighted MRI.
Amide proton transfer weighted MRI | Imaging repeated twice with ~10 weeks between them.
  APT-CEST MRI.
Progression-free survival | Until an event (average 6 months) or closure of the protocol after 4 years.
  Time until progression or death.
Overall survival | Until an event (average 15 months) or closure of the protocol after 4 years.
  Time until death.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared in anonymized form if the local juridical office accepts that full anonymization can be achieved.